CLINICAL TRIAL: NCT06023589
Title: A Multicentre, Randomised, Double-Blind, Parallel-Group Placebo-Controlled, Phase 3, Efficacy and Safety Study of Tezepelumab in 5 to < 12 Year Old Children With Severe Uncontrolled Asthma (HORIZON)
Brief Title: A Study to Investigate the Efficacy and Safety of Tezepelumab Compared With Placebo in Children 5 to < 12 Years Old With Severe Asthma
Acronym: HORIZON
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5180C00016
Record Dates: First submitted 2023-07-20; First posted 2023-09-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Asthma
Keywords: Asthma; Uncontrolled Asthma; Severe Uncontrolled Asthma; Human monoclonal antibody (IgG2λ) cytokine
MeSH Terms: conditions — Asthma | interventions — tezepelumab

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 2:1 ratio to either tezepelumab or matching placebo both administered subcutaneously
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tezepelumab (Experimental): Participants will be receiving tezepelumab subcutaneous injection
  Interventions: Biological: Tezepelumab
- Placebo (Placebo Comparator): Participants will be receiving placebo through a subcutaneous injection
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Tezepelumab — Participants will be receiving subcutaneous injection of tezepelumab
  Other Names: MEDI9929 and AMG157
  Arms: Tezepelumab
Other: Placebo — Participants will be receiving subcutaneous injection of matching placebo
  Arms: Placebo

SUMMARY:
To assess the efficacy and safety of tezepelumab in pediatric participants with severe uncontrolled asthma on medium to high-dose inhaled corticosteroids (ICS) and at least one additional asthma controller medication with or without oral corticosteroids.

DETAILED DESCRIPTION:
This is a phase-3 multicentre, double-blind, parallel-group placebo-controlled, randomised study.

The study will comprise of:

1. Screening/Run-in period of 4 to 6 weeks,
2. 52-week double-blind Treatment period,
3. Post-treatment Follow-up period of 12 weeks.

Participants will be randomised 2:1 to receive either tezepelumab or placebo administered by (SC) Subcutaneous injections for 52 weeks (double-blind Treatment period).

There will then be a 12-week off-treatment Follow-up period for participants who do not continue in the optional open-label Active Treatment Extension period.

An optional open-label Active Treatment Extension will allow all eligible participants the opportunity to receive active treatment with tezepelumab. The Active Treatment Extension period of the study will start following the 52-week double-blind Treatment period and will consist of a 104-week open-label Treatment period prior to the 12-week post-treatment Follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent from (ICF) at least one parent/caregiver (as per local guidelines) and accompanying informed assent from the participant (where the participant is able to provide assent) prior to admission to the study.
2. Participants must be 5 to < 12 years of age, at the time of signing the assent form (as applicable per local guidelines) and their caregivers signing the ICF and at Visit 3.
3. Documented physician diagnosis of severe asthma confirmed and evaluated for at least 6 months prior to Visit 1.
4. Documented physician-prescribed treatment with a total daily dose of either medium or high dose, for at least 3 months with stable dose ≥ 1 month prior to Visit 1.
5. Documented treatment with at least one additional maintenance asthma controller medication is required according to local guidelines and standard of care; (long-acting beta agonist, leukotriene receptor antagonist, long-acting muscarinic antagonist) for at least 3 months with stable dose ≥ 1 month prior to Visit 1.
6. Supportive evidence of asthma as documented by one of the following:

   1. Post-BD (albuterol/salbutamol) responsiveness of FEV1 ≥ 10% during Screening (15 to 30 min after administration of 4 puffs of albuterol/salbutamol with a maximum of 12 puffs of reliever medication only if tolerated by the participant) at either Visit 1 or Visit 2.

      If (a) is not achieved at Visit 1 or Visit 2, historical documentation by any of the below prior to Visit 1:
   2. Post-BD responsiveness of FEV1 ≥ 10%.
   3. Positive methacholine challenge defined as provocative concentration (PC20) of ≤ 16 mg/mL.
   4. PEF average daily diurnal variability > 13% over a 2-week period.
   5. Variability of FEV1 ≥ 12% between any two clinical visits.
   6. Positive exercise challenge test (defined as a fall in FEV1 of > 12%).
   7. FeNO ≥ 20 ppb despite confirmed ICS maintenance therapy.
7. History of at least 2 severe asthma exacerbation events OR 1 severe asthma exacerbation event resulting in hospitalisation within 12 months prior to Visit 1.
8. Pre-BD FEV1 >50% and ≤ 95%PN OR FEV1/forced vital capacity (FVC) ratio ≤ 0.85 at either Visit 1 or Visit 2.
9. Evidence of uncontrolled asthma, with at least 1 of the below criteria:

   1. ACQ-IA score ≥ 1.5 at least once during Screening/Run-in, including Visit 3 (prior to Randomisation) for participants ≥ 6 years old at Screening.
   2. Use of reliever medication, other than as a preventive for exercise induced bronchospasm, on 3 or more days per week for at least 1 week during the Screening/Run-in period.
   3. Sleep awakening due to asthma symptoms requiring use of reliever medication at least once during the Screening/Run-in period.
   4. Asthma symptoms 3 or more days per week in at least 1 week during the Screening/Run-in period.
10. Body weight ≥ 16 kg at Visit 1 (Screening) and Visit 3 (Randomisation).

Exclusion Criteria:

1. History of vocal cord dysfunction, cystic fibrosis, primary ciliary dyskinesia, or chronic rhinosinusitis with nasal polyposis.
2. History of any clinically significant disease or disorder other than asthma which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
3. History of a clinically significant deterioration in asthma or asthma exacerbation including those requiring use of systemic corticosteroids or increase in the maintenance dose of oral corticosteroids within 30 days prior to Visit 1.
4. Change in ICS dose within 1 month prior to Visit 1.
5. History of a life-threatening asthma exacerbation resulting in a hypoxic seizure or requiring intubation.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 231 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2030-08-23 (Estimated)

PRIMARY OUTCOMES:
Annualized severe asthma exacerbation rate (AAER) | From Baseline to Week 52
  To assess the effect of tezepelumab on severe asthma exacerbations in children 5 to < 12 years old with severe uncontrolled asthma compared with placebo.

SECONDARY OUTCOMES:
Change from baseline in pre-bronchodilator (pre-BD) forced expiratory volume in 1 second (FEV1) percent predicted normal (PN) | From Baseline to Week 52
  To assess the effect of tezepelumab on pulmonary function (FEV1) in children with severe uncontrolled asthma compared with placebo. Pre-bronchodilator FEV1% PN will be determined by spirometry at the clinic visit.
AAER associated with allergic asthma | From Baseline to Week 52
  AAER will be assessed in association with both allergic asthma (defined by a positive perennial allergen using serum specific IgE [FEIA]).
Time to first severe asthma exacerbation | From Baseline to Week 52
  Time to first severe asthma exacerbation will be assessed.
Proportion of participants with ≥ 1 severe asthma exacerbation | From Baseline to Week 52
  Proportion of participants with ≥ 1 severe asthma exacerbation will be assessed.
AAER associated with ER visit or hospitalisation | From Baseline to Week 52
  AAER will be assessed in association with ER visits or hospitalisations.
Cumulative exposure to systemic corticosteroids for treatment of severe asthma exacerbations | From Baseline to Week 52
  Cumulative exposure to systemic corticosteroids for treatment of severe asthma exacerbations over the 52 week double-blind treatment period
Change from baseline in Paediatric Asthma Quality of Life Questionnaire (PAQLQ-(S)-IA) total score | From Baseline to Week 52
  Change from baseline of PAQLQ-(S)-IA total score will be assessed. The PAQLQ was developed to measure the functional problems (physical, emotional, and social) that are most troublesome to children with asthma. The PAQLQ-(S)-IA has 23 questions in 3 domains (symptoms, activity limitation, and emotional function). Participants are asked to think about how they have been during the previous week and respond to each question on a 7-point scale (1 = extremely bothered to 7 = not bothered at all or 1 = all of the time to 7 = none of the time). There are 2 coloured cards (green and blue), which list sets of response options appropriate to different questions. The appropriate card should be used by the participant during completion of each question and then taken back when it is no longer required. The overall PAQLQ-(S)-IA score is the mean of all 23 responses, and the individual domain scores are the means of the items in those domains.
Change from baseline in weekly mean daily Paediatric Asthma Symptom Observer (PASO) score | From Baseline to Week 52
  Change from baseline in PASO score will be assessed. The PASO questionnaire will be completed by the caregiver each day from the evening of Treatment period. Caregivers in this study will complete 4 items from the morning assessment capturing night-time asthma symptoms, rescue medication use, night-time awakenings, and maintenance asthma medication use. The evening assessment will capture daytime asthma symptoms, rescue medication use, activity limitation and change in asthma.
Change from baseline in Asthma Control Questionnaire - Interviewer Administered (ACQ-IA) score | From Baseline to Week 52
  Change from baseline in ACQ-IA score will be assessed. The ACQ-IA will only be completed for participants ≥ 6 years old at Screening. The ACQ-IA is administered by trained individuals according to standardised instructions to help the child understand concepts like symptoms (night-time waking, symptoms on waking, activity limitation, shortness of breath, and wheezing) and use of SABA during the past week using a 7-point scale. The ACQ-IA score is calculated by taking the mean of the 6 equally weighted items and ranges from 0 (well controlled) to 6 (extremely poorly controlled). The estimated minimal clinically important difference is 0.5
Change from baseline in weekly mean rescue medication use | From Baseline to Week 52
  Change from baseline in weekly mean rescue medication use will be assessed.
Change from baseline in weekly mean number of night-time awakenings | From Baseline to Week 52
  Change from baseline in weekly mean number of night-time awakenings will be assessed.
Change from baseline in blood eosinophil count | From Baseline to Week 52
  Change from baseline in blood eosinophil count will be assessed.
Change from baseline in fractional exhaled nitric oxide (FeNO) | From Baseline to Week 52
  Change from baseline in FeNO will be assessed.
Change from baseline in total serum IgE | From Baseline to Week 52
  Change from baseline in total serum IgE will be assessed.
Change from baseline in pre-bronchodilator (pre-BD) peak expiratory flow (PEF) | From Baseline to Week 52
  The effect of tezepelumab on pulmonary function compared with placebo will be assessed using spirometry.
Number of asthma--related healthcare resource utilization (HRU) | From Baseline to Week 52
  Mean number and type of Asthma specific HRU (eg, unscheduled physician visits, unscheduled phone calls to physicians, use of other asthma medications) will be assessed.
Number of participant/caregiver health-related absences | From Baseline to Week 52
  Mean number of participant/caregiver health-related absences from work/school due to asthma will be assessed.
Serum concentrations of tezepelumab | At Baseline, Week 4, Week 24, and Week 52
  To evaluate the pharmacokinetics of tezepelumab.
Incidence of anti-drug antibodies (ADAs) | At Baseline, and from time of first dose at Week 0 to end of study at week 64
  To evaluate the immunogenicity of tezepelumab.
Incidence of neutralising antibodies (nAbs) | At Baseline, and from time of first dose at Week 0 to end of study at week 64
  To evaluate the immunogenicity of tezepelumab.

CONTACTS AND LOCATIONS:
Locations (124):
- United States (26):
  - Research Site, Montgomery, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, La Jolla, California
  - Research Site, Long Beach, California
  - Research Site, Orange, California
  - Research Site, San Diego, California
  - Research Site, Atlanta, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Northfield, New Jersey
  - Research Site, Schenectady, New York
  - Research Site, Staten Island, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Columbia, South Carolina
  - Research Site, Coppell, Texas
  - Research Site, Dallas, Texas
  - Research Site, Frisco, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Temple, Texas
- Argentina (8):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Florida
  - Research Site, Lanús
  - Research Site, Lobos
  - Research Site, Mendoza
  - Research Site, Quilmes
  - Research Site, Rosario
- Brazil (5):
  - Research Site, Blumenau
  - Research Site, Curitiba
  - Research Site, Salvador
  - Research Site, São Paulo
  - Research Site, Sorocaba
- Canada (5):
  - Research Site, Edmonton, Alberta
  - Research Site, Burlington, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Montreal, Quebec
- China (8):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Lanzhou
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Wuxi
- Colombia (2):
  - Research Site, Bogotá
  - Research Site, Medellín
- France (7):
  - Research Site, Brest
  - Research Site, Bron
  - Research Site, Créteil
  - Research Site, Marseille
  - Research Site, Paris
  - Research Site, Rouen
  - Research Site, Vandœuvre-lès-Nancy
- Hungary (3):
  - Research Site, Debrecen
  - Research Site, Szeged
  - Research Site, Szigetvár
- Italy (3):
  - Research Site, Genova
  - Research Site, Pavia
  - Research Site, Roma
- Japan (9):
  - Research Site, Fukuoka
  - Research Site, Fukuyama
  - Research Site, Funabashi-shi
  - Research Site, Nara
  - Research Site, Odawara
  - Research Site, Ōtsu
  - Research Site, Saga
  - Research Site, Shimotsuga-gun
  - Research Site, Yokohama
- Mexico (4):
  - Research Site, Chihuahua City
  - Research Site, Guadalajara
  - Research Site, Mexico City
  - Research Site, Veracruz
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Rotterdam
- Philippines (4):
  - Research Site, Iloilo City
  - Research Site, Las Piñas
  - Research Site, Quezon
  - Research Site, Santa Rosa
- Poland (2):
  - Research Site, Lodz
  - Research Site, Tarnów
- Research Site, Bucharest, Romania
- South Africa (7):
  - Research Site, Bellville
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Middelburg
  - Research Site, Thabazimbi
  - Research Site, Vereeniging
  - Research Site, Welkom
- South Korea (2):
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (7):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Esplugues de Llobregat (Barc)
  - Research Site, Madrid
  - Research Site, Sabadell
  - Research Site, Valencia
  - Research Site, Villarreal
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Bangkoknoi
  - Research Site, Chiang Mai
  - Research Site, Muang
- Turkey (Türkiye) (4):
  - Research Site, Bursa
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Yenimahalle
- Ukraine (3):
  - Research Site, Chernivtsi
  - Research Site, Ivano-Frankivsk
  - Research Site, Kyiv
- United Kingdom (8):
  - Research Site, Birmingham
  - Research Site, Bradford
  - Research Site, Bristol
  - Research Site, Glasgow
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Nottingham
  - Research Site, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/